CLINICAL TRIAL: NCT05602428
Title: Traditional Chinese Medicine Hospital of Changzhou Affiliated to Nanjing University of Traditional Chinese Medicine
Brief Title: Analysis of Clinical Effect of Subanesthetic Dose of Esketamine Combined With Hip Capsule Peripheral Nerve Block in Elderly Patients Undergoing Total Hip Arthroplasty
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Changzhou Traditional Chinese Medicine Hospital Affiliated to Nanjing University of Chinese Medicine (Other)
Responsible Party: Principal Investigator, Yanhua Huo, Doctor, Changzhou Traditional Chinese Medicine Hospital Affiliated to Nanjing University of Chinese Medicine
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: ChangzhouTCMH
Record Dates: First submitted 2022-09-20; First posted 2022-11-02 (Actual); Last update posted 2022-11-02 (Actual); Status verified 2022-10

CONDITIONS: Total Hip Arthroplasty

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- The observation group A (Experimental): The use of esketamine sub-anesthetic dose combined with hip capsule peripheral nerve block. The patients were subjected to local anesthesia and punctured through the left radial artery for invasive arterial blood pressure monitoring. Anesthesia induction: the observation group followed by intravenous injection of ketamine 0.2mg/kg, sufentanil 0.3μg/kg, Cyclophenol 0.3mg/kg, midazolam 2mg, rocuronium 0.6mg/kg. After the onset of the drug endotracheal intubation, connect anesthesia machine control breathing. Anesthesia was maintained with 1%~2% sevoflurane inhalation, remifentanil infusion rate was 0.2~0.3 μg/kg·min, sevoflurane was stopped 30 min before the end of the operation. Patient-controlled intravenous analgesia pump (PCIA) was given for postoperative analgesia. PCIA formula: sufentanil 100ug+ondansetron 8mg+ketorolac tromethamine 60mg+saline to 100ml, pump speed 2ml/h, automatic single dose 3ml, lock time 20min.
  Interventions: Drug: esketamine sub-anesthetic,
- the control group B (Active Comparator): Esketamine subanesthetic dose combined with lumbar plexus block was used. The patient was placed in the healthy lateral decubitus position and ultrasound-guided puncture was performed 4 cm beside the 3rd and 4th lumbar vertebrae (Figure 1B、C). The frequency of the ultrasound probe was 2-5 MHz, and the probe was adjusted until the images below the transverse processes of the 3rd to 5th lumbar vertebrae and the psoas muscle were clearly displayed, and the needle was inserted close to the probe and retracted in the lumbar plexus, and sufentanil 0.5 μg/kg, propofol 1.5 mg/kg, and rocuronium 0.6 mg/kg were injected after no blood extraction. General anesthesia was then performed using a subanesthetic dose of esketamine and the same maintenance and postoperative analgesic measures were used as in group A.
  Interventions: Drug: esketamine sub-anesthetic
- the control group C (Active Comparator): general anesthesia was performed with esketamine subanesthetic dose. The same maintenance and postoperative analgesia measures were used as in group A.
  Interventions: Drug: esketamine sub-anesthetic

INTERVENTIONS:
Drug: esketamine sub-anesthetic, — the use of esketamine sub-anesthetic dose combined with hip capsule peripheral nerve block
  Arms: The observation group A
Drug: esketamine sub-anesthetic — Esketamine subanesthetic dose combined with lumbar plexus block was used
  Arms: the control group B
Drug: esketamine sub-anesthetic — general anesthesia was performed with esketamine subanesthetic dose.
  Arms: the control group C

SUMMARY:
To observe the clinical effect of esketamine combined with hip capsule peripheral nerve block in elderly patients undergoing total hip arthroplasty. A total of 120 elderly patients who underwent total hip arthroplasty in our hospital from January 2020 to May 2021 were randomly divided into three groups, 40 cases in each group. The observation group A was treated with esketamine subanesthetic dose combined with hip capsule peripheral nerve block, the control group B was treated with esketamine subanesthetic dose combined with lumbar plexus block, and the control group C was treated with esketamine subanesthetic dose for general anesthesia. The onset time of anesthesia, duration of block, postoperative recovery time, postoperative extubation time, MAP and HR indexes before anesthesia (T0), during skin incision (T1), 30 minutes after the start of surgery (T2), and at the end of surgery (T3) were recorded in the three groups, and the VAS score and Ramsay score at 0.5 h, 2 h, 6 h, 12 h, and 24 h after surgery, as well as the incidence of postoperative adverse reactions were recorded in the three groups.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged ≥ 60 years
* American Society of Anesthesiology (ASA) II or III
* No serious coronary heart disease, hypertension, diabetes and related complications, no serious liver and kidney function damage, no mental illness

Exclusion Criteria:

* Allergic to ketamine
* Abnormal coagulation function
* Mental system diseases or cognitive dysfunction
* Severe liver and kidney dysfunction

Min Age: 60 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Actual)
Dates: Start 2020-01-01 (Actual); Primary Completion 2021-05-31 (Actual); Study Completion 2021-05-31 (Actual)

PRIMARY OUTCOMES:
Anesthesia indicators | onset time of anesthesia 5 minutes
  Add a onset time of anesthesia Outcome Measure
Anesthesia indicators | duration of block time 350 minutes
  Add a duration of block Outcome Measure
Anesthesia indicators | postoperative recovery time 15 minutes
  Add a postoperative recovery time Outcome Measure
Anesthesia indicators | postoperative extubation time 17 minutes
  Add a postoperative extubation time Outcome Measure
Vital signs | before anesthesia (T0)
  mean arterial pressure before anesthesia (T0)
Vital signs | during skin incision (T1)
  mean arterial pressure during skin incision (T1)
Vital signs | 30 minutes after the start of surgery (T2)
  mean arterial pressure 30 minutes after the start of surgery (T2)
Vital signs | at the end of surgery (T3) 85 minutes
  mean arterial pressure at the end of surgery (T3)
Vital signs | before anesthesia (T0)
  heart rate before anesthesia (T0)
Vital signs | during skin incision (T1)
  heart rate 30 minutes during skin incision (T1)
Vital signs | after the start of surgery (T2)
  heart rate after the start of surgery (T2)
Vital signs | at the end of surgery (T3) 78 minutes
  heart rate at the end of surgery (T3)
Visual Analogue Scale | 0.5hour
  Visual Analogue Scale score (0 is no pain; 0 ~ 4 is mild pain; 4 ~ 7 is moderate pain; 7 ~ 10 is severe pain)
Visual Analogue Scale | 2hour
  Visual Analogue Scale score (0 is no pain; 0 ~ 4 is mild pain; 4 ~ 7 is moderate pain; 7 ~ 10 is severe pain)
Visual Analogue Scale | 6hour
  Visual Analogue Scale score (0 is no pain; 0 ~ 4 is mild pain; 4 ~ 7 is moderate pain; 7 ~ 10 is severe pain)
Visual Analogue Scale | 12hour
  Visual Analogue Scale score (0 is no pain; 0 ~ 4 is mild pain; 4 ~ 7 is moderate pain; 7 ~ 10 is severe pain)
Visual Analogue Scale | 24hour
  Visual Analogue Scale score (0 is no pain; 0 ~ 4 is mild pain; 4 ~ 7 is moderate pain; 7 ~ 10 is severe pain)
Ramsay sedation score | 0.5hour
  Ramsay score (range 0~6 points, 1 point for insufficient sedation, 2~4 points for good sedation, 5~6 points for excessive sedation)
Ramsay sedation score | 2hour
  Ramsay score (range 0~6 points, 1 point for insufficient sedation, 2~4 points for good sedation, 5~6 points for excessive sedation)
Ramsay sedation score | 6hour
  Ramsay score (range 0~6 points, 1 point for insufficient sedation, 2~4 points for good sedation, 5~6 points for excessive sedation)
Ramsay sedation score | 12hour
  Ramsay score (range 0~6 points, 1 point for insufficient sedation, 2~4 points for good sedation, 5~6 points for excessive sedation)
Ramsay sedation score | 24hour
  Ramsay score (range 0~6 points, 1 point for insufficient sedation, 2~4 points for good sedation, 5~6 points for excessive sedation)
Adverse reactions | at the end of surgery 48 hours
  the incidence of postoperative delirium, nausea and vomiting, drowsiness, skin itching and other adverse reactions

CONTACTS AND LOCATIONS:
Overall Officials: Yanhua Huo, BM, Principal Investigator — Traditional Chinese Medicine Hospital of Changzhou Affiliated to Nanjing University of Traditional Chinese Medicine
Locations (1):
- ChangzhouTCMH, Changzhou, Jiangsu, China

IPD SHARING:
Plan to Share IPD: Undecided